CLINICAL TRIAL: NCT03374904
Title: Video Feedback Intervention to Enhance Parental Reflective Function in Primary Caregivers of Children With Severe Psychiatric Disorders. Feasibility Randomized Trial
Brief Title: Video Feedback to Enhance Parental Mentalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Valparaiso (Other)
Collaborators: Pontificia Universidad Catolica de Chile (Other); University of Chile (Other)
Responsible Party: Principal Investigator, Fanny Leyton, Psychiatrist at Child Inpatient Unit, Principal Investigator, Universidad de Valparaiso
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0020173081
Record Dates: First submitted 2017-10-19; First posted 2017-12-15 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Parenting
Keywords: Parenting; Parental Mentalization; Parental Reflective Function; Child Psychopathology
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to intervention or control group at a 2:1 ratio
Who Masked: Outcomes Assessor
Masking Description: Interview analysis, for ascertaining the level of PRF will be done by an encoder highly trained in said techniques. Transcriptions will be anonymous in order to mask the identity of the caregiver. Whether the caregiver belongs to a control or intervened group will also be masked when working in transcriptions.
  Due to the characteristics of the intervention, the main researcher will not be masked regarding who receives the intervention and who is in the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Patients in control group will attend to four session of Play Therapy plus inpatient treatment as usual during four weeks
  Interventions: Behavioral: Control Group
- Video Feedback (Experimental): Once a week, after play therapy, individual or group video feedback session will be done.
  Interventions: Behavioral: Video Feedback; Behavioral: Control Group

INTERVENTIONS:
Behavioral: Video Feedback — first, a play interaction between the child and caregiver is recorded (5 to 10 minutes), then the therapist and caregivers watch together a selected part of the video (1 to 2 minutes) and provide feedback with a six step protocol.
  Other Names: Video Intervention Therapy
  Arms: Video Feedback
Behavioral: Control Group — Play therapy will be administered once a week plus inpatient treatment as usual for 4 weeks
  Other Names: Treatment us Usual

SUMMARY:
The objective of this study is to implement a Video Feedback (VF) intervention to enhance Parental Reflective Function in primary caregivers of inpatient psychiatric children. Because there is no published research using VF with parents of children with severe psychopathology and in hospitalized context, this study is a pilot study.

The research will include a qualitative and quantitative study; it will take place in a public hospital in Valparaíso, Chile. In the qualitative study, participants will be six primary caregivers who received the intervention and three stakeholders from Child Unit. For caregivers a semi-structured interview will be applied to know subjective experience gained by intervention regarding the perceived satisfaction. For health professional also a semi-structured interview will be applied to collect information pertinent to the feasibility of performing such intervention. The information obtained from the interviews will be analyzed with Grounded Theory model.

The quantitative study will be conducted amongst all tutors of children aged between 6 and 14 hospitalized in a child psychiatry ward between August 2017 and December 2018. The expected sample size is 30 subjects in total; 10 for the control group and 20 for the experimental group.

A four module of Video Intervention Therapy (VIT) was designed, each module includes a (video recorded) play session and a group VF session.

The evaluation of the caregivers at the beginning of the intervention will include a psychosocial questionnaire, GHQ-12 , Five Minutes Speech Sample (FMSS) where RF will be codified, Operationalized Psychodynamic Diagnosis - Structure Questionnaire (OPD.SQ). The Strengths and Difficulties Questionnaire will be applied to children, in addition to the Children Global Assessment Scale, (CGAS). After every VF session a new FMSS, GHQ-12 and CGAS will be made. A follow-up will be performed three months after the beginning of the intervention with FMSS, GHQ-12 for caregivers and SDQ and CGAS for children.

To determine Effect Size and Intra Class Correlation, the results will be analyzed using a multiple linear regression.

DETAILED DESCRIPTION:
One of the challenges when a child is hospitalized is working with the family, there is an enormous evidence relating family factors with onset of psychopathology and pour outcomes in children. Usually treatment includes parental support or family therapy, but most parents attend to few sessions.

Mentalization is defined as the capacity to understand and interpret one's own behavior and those of others as an expression of mental states, such as feelings, thoughts, fantasies, beliefs and desires. Reflective function (RF) is the operational definition of mentalization. Parental mentalizing is considered to have important implications for the development of self-regulation in Children.

Video assisted therapy has demonstrated to be a powerful tool in promoting change in parent-child relationships with few sessions.

The present study

To assess a short program aimed at improving Parental Reflective Function (PRF) during the hospitalization of children and early adolescents admitted to a psychiatric unit, a randomized pilot psychotherapeutic intervention using video feedback has been designed as a clinical trial. There is ample evidence of the usefulness of video feedback to increase sensitivity and PRF in children up to 5 years, but in older children the evidence is limited. There are no known published randomized clinical trials using video feedback in parents of children admitted for psychiatric reasons.

A VF therapy like this will allow implementing a short and economic intervention, which has been used in older children and in parents with mental health problems, as is expected in parents of inpatient psychiatric children. This research also will contribute to explore how PRF relates to children psychopathology.

General objectives

1. To assess the feasibility and acceptability of a psychotherapeutic intervention using video feedback in order to improve the PRF in primary caregivers of children and adolescents hospitalized in public inpatient unit.
2. To provide data to estimate the parameters required to design a definitive Randomized Control Trial with a psychotherapeutic intervention using VF in order to improve the PRF in primary caregivers of children and adolescents hospitalized in public inpatient unit.

Method This project was approved by the Ethics Committee of the Valparaíso-San Antonio Health Service The research has the support of the head of the Child Psychiatry Unit and the Director of the Psychiatric Hospital.

Participants The research will take place in a public child/adolescent psychiatry ward in Valparaíso in "Hospital Psiquiátrico del Salvador"

In the qualitative study, participants will be a minimum of six primary caregivers of children hospitalized in a psychiatric ward receiving intervention between the ages of 6 and 14, as well as three key players (a therapist, a nurse and chief psychiatrist of the Special Care Unit).

The quantitative study will be conducted amongst all tutors of children hospitalized in a child psychiatry ward between August 2017 and December 2018. The sample will be all parents and/or caregivers that meet the inclusion criteria and wish to participate. The expected sample size is 30 subjects in total; 10 for the control group and 20 for the experimental group. If by December 2018 the total sample has not been met, more subjects will be recruited in order to achieve the sample size. A clinical essay having 30 subjects has been proposed because an intervention of these characteristics has not been performed in Chile; so the impact of the effect must first be estimated in order to assess the feasibility for a future multi-centric clinical trail. This is the reason behind piloting the present study.

Procedure

Qualitative study. Two semi-structured interview scripts will be performed.

* One script aims to gain full grasp of the subjective experience gained by intervention participants regarding the perceived workshop satisfaction and follow-up.
* The second script will be aimed at key institutional information holders, aiming to collect information pertinent to the feasibility of performing such an intervention. Questions will focus on analyzing the necessary resources needed and impact the workshop may have in the functioning of the child psychiatric ward.

The interviews will be performed by physicians undergoing a psychiatrist specialization and/or a psychologist who is not participating in the intervention.

Quantitative Study

At the onset of hospitalization, all caregivers meeting inclusion criteria must provide an informed consent form in order to participate in the study. Children must provide an informed approval after caregivers have provided their consent.

All caregivers that participate in the study will receive an array of instruments upon entering, subsequently randomized between the control groups and those intervened. If any mental health problem is detected in caregivers it will be made a referral for her or him to get special support according to the problem detected

Both groups of caregivers along with their child receive the same regular care and treatments they would normally receive from a inpatient unit. Since both groups will be subject to a larger intervention, the aim of a future randomized control trial will be to objectify how much VF boosts the improvement of PRF during a child's psychiatric hospitalization.

Intervention Interventions will be performed by the principal investigator and by a child clinical psychologist, both trained and supervised in Video Intervention Therapy (VIT). VIT is a technique for performing Video Feedback where behavior-oriented interventions and representational therapy elements are used. This provides a six-step video analysis framework. The video may be filmed at different settings, the only requirement being a visual interaction of the child with his parents.

A four module intervention was designed for this study, each module includes a play session and a VF session. The play session has a workshop format, it has a duration of 45 to 60 minutes, where the caregiver(s) plays freely with the child. During the play session, a five to ten minute video sessions of the dyads will be made. The therapeutic team will then pick approximately 1 minute long excerpts to display in the VF sessions. The VF sessions will occur during the same week and these could be group sessions.

Analysis plan

Qualitative Study The information obtained from the interviews will be analyzed with Grounded Theory model, obtained open codify data.

For the analysis the ATLAS.TI Software will be used, enabling managing and processing text data groups.

Quantitative Study

1. A descriptive statistic will be performed to compare the control group and the intervened group regarding clinical and sociodemographic variables.
2. It will be also presenting descriptive statistic on eligibility rate, recruitment rate, and compliance.
3. To determine Effect Size and Intra Class Correlation results will be analyzed using a multiple linear regression, multi level model with randomized and fixed interception.

Quantitative data will be analyzed using STATA 14.

ELIGIBILITY:
Inclusion Criteria:

* Figure as a tutor during hospitalization or,
* Figure as the primary caregiver of the child or adolescent and,
* Must have a (legal or biological) kinship with the hospitalized child or adolescent.

Exclusion Criteria:

* Responsible adults that present a severe intellectual deficit or psychotic symptoms or,
* Institutional caregivers or,
* Parents that do not care for the child regularly (see the child lees than a week per month, has restraining orders, etc. )

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-04-23 (Actual)

PRIMARY OUTCOMES:
Feasibility of delivering the intervention | Through study completion, approximately 18 months
  Estimate the proportion of the quantity of performed sessions against the quantity of planned VF sessions.
Feasibility as measured by participant retention | Through study completion, approximately 21 months
  Number of participants who remain in the study at the 12 weeks follow up
Feasibility of recruitment | Through study completion, approximately 18 months
  Estimate the proportion of caregivers who meet eligibility criteria and accept the invitation to participate in the study (recruiting rate)
Acceptability as measured by compliance-to-intervention rate | Through study completion, approximately 18 months
  proportion of caregivers that complete the intervention against the quantity of randomized.
Change over time in Caregiver's Parental Reflective Function | Baseline (T0), weekly during 4 weeks after allocation (T1, T2, T3, T4) and 12 weeks follow up (T5)
  Parental Reflective Function is obtained from a general codification of the Five Minutes Speech Sample transcription according to the Reflexive Function Evaluation Manual with a scale that goes from -1 (avoidance or rejection of the mentalization) to 9 score points (complete or exceptional RF). A score of 5 reflects a clear understanding of mental states.

SECONDARY OUTCOMES:
Acceptability of the intervention by primary caregivers | Following completion of the intervention (4 weeks from allocation)
  Satisfaction and related factors from the caregivers perspective that participate in the VF intervention, it will be assessed through a qualitative semi-structured interview
Acceptability of the intervention by key stakeholders (a therapist, a psychiatrist and a nurse) of child inpatient unit | Through study completion, approximately 21 months
  Acceptability of performing a novel intervention from health professionals it will be assessed through a qualitative semi-structured interview.
Operationalized Psychodynamic Diagnosis - Structure Questionnaire (OPD-SQ) 12 item version | Baseline (T0)
  OPD-SQ Auto report instrument that measures the level of structural integration of personality in 12 items, in which people indicate the degree to which they feel accurately described in a 5 point Likert scale. Higher scores are indicators of less structural integration.
Change over time The General Health Questionnaire (GHQ-12) in Caregivers | Baseline (T0), weekly during 4 weeks after allocation (T1, T2, T3, T4) and 12 weeks follow up (T5)
  The well-being of parents will be measured using a 12-question questionnaire to measure overall psychological well-being. Total scores range from 0 to 36. Higher scores indicate more psychological problems
Change over time in Strengths and Difficulties Questionnaire (SDQ) in Children | Baseline (T0), weekly during 4 weeks after allocation (T1, T2, T3, T4) and 12 weeks follow up (T5)
  The parents' self-reported behavior using the Strengths and Difficulties Questionnaire (SDQ), a 25-item questionnaire that assesses children's positive and negative attributes, each item uses a 3-point Likert ordinal scale. The answers have a score of 0-2 for the items written negatively and a reverse score of 2-0 for the items written positively. Thus, higher scores indicate more problematic attributes for all the 25 items
Change over time in Clinical Global Impression Scale (CGAS) in Children | Baseline (T0), weekly during 4 weeks after allocation (T1, T2, T3, T4) and 12 weeks follow up (T5)
  Change in Severity of Psychopathology with Clinical Global Impression Scale (CGAS),

CONTACTS AND LOCATIONS:
Overall Officials: Fanny Leyton, Md, Principal Investigator — Hospital Psiquiátrico del Salvador. Universidad de Valparaíso
Locations (1):
- Hospital Psiquiátrico del Salvador, Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bakermans-Kranenburg MJ, van IJzendoorn MH, Juffer F. Less is more: meta-analyses of sensitivity and attachment interventions in early childhood. Psychol Bull. 2003 Mar;129(2):195-215. doi: 10.1037/0033-2909.129.2.195. PMID 12696839
- [Background] Beebe B. Mother-infant research informs mother-infant treatment. Psychoanal Study Child. 2005;60:7-46. doi: 10.1080/00797308.2005.11800745. PMID 16649674
- [Background] Benbassat N, Priel B. Parenting and adolescent adjustment: the role of parental reflective function. J Adolesc. 2012 Feb;35(1):163-74. doi: 10.1016/j.adolescence.2011.03.004. Epub 2011 Apr 16. PMID 21497896
- [Background] Fukkink RG. Video feedback in widescreen: a meta-analysis of family programs. Clin Psychol Rev. 2008 Jul;28(6):904-16. doi: 10.1016/j.cpr.2008.01.003. Epub 2008 Feb 5. PMID 18359136
- [Background] Shaffer D, Gould MS, Brasic J, Ambrosini P, Fisher P, Bird H, Aluwahlia S. A children's global assessment scale (CGAS). Arch Gen Psychiatry. 1983 Nov;40(11):1228-31. doi: 10.1001/archpsyc.1983.01790100074010. PMID 6639293
- [Background] Steele M, Steele H, Bate J, Knafo H, Kinsey M, Bonuck K, Meisner P, Murphy A. Looking from the outside in: the use of video in attachment-based interventions. Attach Hum Dev. 2014;16(4):402-15. doi: 10.1080/14616734.2014.912491. PMID 24972107
- [Background] Facchini S, Martin V, Downing G. Pediatricians, Well-Baby Visits, and Video Intervention Therapy: Feasibility of a Video-Feedback Infant Mental Health Support Intervention in a Pediatric Primary Health Care Setting. Front Psychol. 2016 Feb 16;7:179. doi: 10.3389/fpsyg.2016.00179. eCollection 2016. PMID 26909063
- [Background] Fonagy P, Target M. Bridging the transmission gap: an end to an important mystery of attachment research? Attach Hum Dev. 2005 Sep;7(3):333-43. doi: 10.1080/14616730500269278. PMID 16210243
- [Background] Ortuno-Sierra J, Aritio-Solana R, Fonseca-Pedrero E. Mental health difficulties in children and adolescents: The study of the SDQ in the Spanish National Health Survey 2011-2012. Psychiatry Res. 2018 Jan;259:236-242. doi: 10.1016/j.psychres.2017.10.025. Epub 2017 Oct 18. PMID 29091822
- [Background] Camoirano A. Mentalizing Makes Parenting Work: A Review about Parental Reflective Functioning and Clinical Interventions to Improve It. Front Psychol. 2017 Jan 20;8:14. doi: 10.3389/fpsyg.2017.00014. eCollection 2017. PMID 28163690
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. Pilot Feasibility Stud. 2016 Oct 21;2:64. doi: 10.1186/s40814-016-0105-8. eCollection 2016. PMID 27965879
- [Background] Setoya Y, Saito K, Kasahara M, Watanabe K, Kodaira M, Usami M. Evaluating outcomes of the child and adolescent psychiatric unit: A prospective study. Int J Ment Health Syst. 2011 Mar 31;5:7. doi: 10.1186/1752-4458-5-7. PMID 21453481
- [Derived] Leyton F, Olhaberry M, Moran J, De la Cerda C, Leon MJ, Sieverson C, Alfaro A, Hernandez C, Alvardo R, Steele H. Video Intervention Therapy for primary caregivers in a child psychiatry unit: a randomized feasibility trial. Trials. 2021 Oct 30;22(1):754. doi: 10.1186/s13063-021-05668-w. PMID 34717750
- [Derived] Leyton F, Olhaberry M, Alvarado R, Rojas G, Duenas LA, Downing G, Steele H. Video feedback intervention to enhance parental reflective functioning in primary caregivers of inpatient psychiatric children: protocol for a randomized feasibility trial. Trials. 2019 May 14;20(1):268. doi: 10.1186/s13063-019-3310-y. PMID 31088531